CLINICAL TRIAL: NCT03325699
Title: Support Monitoring and Reminder Technology for Mild Dementia
Brief Title: Support Monitoring and Reminder Technology
Acronym: SMART4MD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johan Sanmartin Berglund (Other)
Collaborators: HealthBit (Unknown); Andaluz Health Service (Other Government); Blekinge Institute of Technology (Other); Consorci Sanitari de Terrassa (Other); DEX Innovation Centre (Unknown); Anglia Ruskin University (Other); University College Leuven - Limburg (Unknown); Universidad Politecnica de Madrid (Other); Athena ICT (Unknown)
Responsible Party: Sponsor-Investigator, Johan Sanmartin Berglund, Professor, MD, PhD, Blekinge Institute of Technology
Organization: Blekinge Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 643399
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Mild Dementia; Cognitive Impairment, Mild
Keywords: Mild dementia; Cognitive impairment; Informal caregiver; Aging; Quality of life; Health application; Information and communication technology (ICT)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants assigned to the intervention group will have access to the SMART4MD health application and participate in clinical visits every 6 months
  Interventions: Device: SMART4MD Health Application
- Control (No Intervention): Participants assigned to the intervention group will NOT have access to the SMART4MD health application and participate in clinical visits every 6 months

INTERVENTIONS:
Device: SMART4MD Health Application — SMART4MD is a general health application which has been adapted specifically for people with mild dementia through a structured process. The application is intended to be used daily at home, mainly by the participants themselves, with the help of their informal carers. The application is optimized for tablet devices running on Android operating system (OS). Participants will be provided with a tablet with the SMART4MD health application.
  The core functionalities of the application are based on reminders (medication, appointments with healthcare providers), brain supporting activities (clock, calendar, brain games, photos) and optional status and health information sharing with family and informal carers (including daily feeling status, specific health problems, and quality of life). An important feature of SMART4MD is its personalization facility: main users (PWD and informal carers) will be able to switch off/on various features and information sharing possibilities.
  Arms: Intervention

SUMMARY:
This multicentre randomized control trial aims to evaluate the effects of an intervention consisting of an health application developed to improve the quality of life (QoL) in older people with mild dementia and their informal caregivers. The study is a collaboration between five European countries where the clinical trials will be conducted in four of these countries (Sweden, Belgium, Spain and Czech Republic).

In total 1200 dyads (consisting of a person with mild dementia (PWD) and their informal caregiver (carer) will be recruited for this study. Participant dyads will be randomized in a 1:1 ratio in two parallel groups: PWD to receive either usual care from primary or specialized providers (control group) or to receive usual care plus access to a tablet with the SMART4MD health application (intervention group).

Participants in the trial will be assessed for a period of 18 months. After the baseline visit, all participants will have follow-up visits every 6 months together with a checkup of the PWDs capacity to remain in the study. In the follow up visits, investigators will assess the PWD's quality of life, their cognitive and functional status, adherence to prescribed medication and attendance at healthcare appointments and admissions to healthcare services institutions. Investigators will also assess the burden of the informal caregivers.

DETAILED DESCRIPTION:
SMART4MD has been developed from an existing general health management application in a process involving the structured participation of PWD, their informal carers, and clinicians.

STANDARD OPERATING PROCEDURES

Participants will be recruited over a period of six months by the nominated/approved licensed providers of relevant medical care at the different sites. Participants will not receive financial reimbursement for taking part in this trial.

Participants will be identified from people with cognitive impairment that has been present for more than six months and who meet all the study eligibility criteria (listed in section Eligibility). The Mini-Mental State Examination (MMSE) and Geriatric Depression Scale (GDS-15) will be used to screen PWD at recruitment. participants can be under primary care services as well as secondary care services. Participants will also be identified from patient databases such as those integrated in the network of Consorci Sanitari de Terrassa (CST) and Database of all patients participating in the Swedish National Study on Aging and Care (SNAC). In order to assure that all clinical sites have a similar approach in recruiting participants, a guide with best practices for patient recruitment have been developed.

The following data will be collected in this trial:

* Mini Mental State examination (MMSE)
* Geriatric Depression Scale (GDS)
* Demographic data
* Medical history - PWD only
* Familiarity with comparable technological devices
* Quality of Life AD (QoL-AD)
* Adherence to medication
* The Lawton Instrumental Activities of Daily Living (IADL)
* EuroQoL 5 Dimension (EQ5D)
* The Short-form Zarit Caregiver Burden Interview (ZBI-12)
* Attendance at healthcare appointments and admissions to healthcare institutions
* Data from the SMART4MD application focusing on user behaviour and usage of core functionalities.

All variables collected in this study is listed and detailed described in a electronic case report form, with associated guidelines, to ensure consistency in all gathered data.

Any relevant changes to physical health will be noted during these investigations including whether the PWD is still in charge of their own medication and whether the same individual is still the informal carer of PWD. In case of an adverse event (AE) or serious adverse event (SAE), medical or psychosocial, the investigator and his or her team are responsible for detecting, recording, reporting and taking appropriate actions in according to the requirements of the local institutional review board (IRB) and the appropriate regulatory body with health- and social care in respective country of the study. Reporting of any AE and SAE must be done within 24 hours by an SAE Report Form sent to the clinical lead of this study.

SAMPLE SIZE ASSESSMENT To compare two groups (Intervention and Control) using a two- sample, two-sided t-test with a 5% statistical significance level, the minimum number of evaluable PWDs required in each group is 470 (940 overall), to give a power of 80%. If there would be a drop-out rate of 20% of the PWDs then the number of PWDs registered on the study would need to be 564 in each group (1128 overall).

STATISTICS ANALYSIS PLAN Data collected for the study will be analyzed to measure and assess the SMART4MD health application impact on QoL-AD for the PWDs as the primary outcome. In addition, functional status (IADL) for PWD, adherence to prescribed medication, health care appointment and admissions records and carer burden will be analyzed as secondary outcome.

All the baseline data variables collected will be summarized by group and overall, and also by site. Among the statistical summary statistics considered for presentation for continuous measures in summary tables will be the mean, median, minima and maxima, lower and upper quartiles, and standard deviation. Categorical variables will be summarized using counts and percentages. As the PWDs will be assigned to the intervention and control using random allocation it is known in advance that any differences between these groups at baseline will be as a result of chance and so no formal comparison of the groups using statistical significance tests will be carried out at baseline.

Primary outcome analysis:

The primary analysis will be the comparison of the 18-month total QoL-AD score means using a two- sample, two-sided Monte Carlo permutation t-test. The use of a permutation test will avoid the need for strong assumptions about the distribution of the data. Similarly, a bootstrap approach will be used to obtain the 95% confidence limits for the difference between the group means.

Secondary outcome analyses:

The secondary analysis focus on a cost-effectiveness and/or cost-utility analysis from a Health Service perspective (financer perspective) measured by QUALYs. Furthermore, a user-behavior analysis of the SMART4MD health application by analyzing the frequency of access to the application, the length of this interaction, and the quality of the inputs provided. Usability tests will be performed based on the System Usability Scale (SUS). At last, a technical familiarity score is calculated to assess prior experience of technology and the effect on the outcomes analyzed by statistical regression analysis.

PLAN FOR MISSING DATA Each partner are responsible for ensuring that any missing data will be reported as missing in the study database.For analyses involving multiple regression analysis a multiple imputation approach will be considered and used if statistically sound, depending on the proportion and pattern of missing values.

QUALITY ASSURANCE PLAN

The monitor(s) will review and report process during the course of the trial covering participant enrolment, consent, eligibility and allocation to trial groups, policies to protect participants, including reporting of harm and completeness, accuracy and timeliness of data collection.

ELIGIBILITY:
Inclusion criteria (PWD only):

* Participants score 20-26 points on Mini-Mental State Examination (MMSE) Participants +55 years of age
* Male or female. No preference will be given to either
* Participants are home-care recipients
* Participants have an informal carer
* Those participants who take prescribed medication are in charge of their own medication use
* Participants have no specific conditions reducing their physical ability to use the application to a point that makes their participation in the project impossible, as evaluated by the responsible investigator (the nature of the conditions should be recorded in such cases)
* The place where the participant is normally resident has sufficient wireless or phone network connectivity to enable them to use SMART4MD on a daily basis
* Cognitive impairment must have been present for more than six months

Exclusion criteria (PWD only):

* Participants have a terminal illness with <3 years expected survival
* Participants score above 11 on the Geriatric Depression Scale (GDS-15)

Ages: 55 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2016-12-03 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Health Related Quality of Life (HRQL) QoL-AD questionnaire (Thorgrimsen et al. 2003; Rebecca G. Logsdon et al. 2002; R. G. Logsdon et al. 1999) | 18 months
  This is a 13-item measure which has been specifically designed to measure QoL in individuals with dementia from the perspective of both the PWD and the informal carer. QoL-AD will be assessed via an interview with PWD and via self-completion by informal carers.

SECONDARY OUTCOMES:
Adherence to medication | 18 months
  Increase adherence to prescribed medication prescription
Mini mental state examination (MMSE) | 18 months
  Reduce functional decline of PWD
Attendance to health care appointments | 18 months
  Monitor PWD´s attendance at health care appointments and admissions to health care institutions
Zarit Burden Interview (ZBI) | 18 months
  Monitor the mental well-being of informal caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Tomer Regev, PhD, Study Director — Anglia Ruskin University
Locations (5):
- University College Leuven - Limburg, Genk, Belgium
- DEX Innovation Centre, Prague, Czechia
- Spain (2):
  - Consorci Sanitaria de Terrassa, Terrassa, Barcelona
  - Servicio Andaluz Salud, Seville
- Blekinge Institute of Technology, Karlskrona, Blekinge County, Sweden

REFERENCES:
- [Derived] Guzman-Parra J, Barnestein-Fonseca P, Guerrero-Pertinez G, Anderberg P, Jimenez-Fernandez L, Valero-Moreno E, Goodman-Casanova JM, Cuesta-Vargas A, Garolera M, Quintana M, Garcia-Betances RI, Lemmens E, Sanmartin Berglund J, Mayoral-Cleries F. Attitudes and Use of Information and Communication Technologies in Older Adults With Mild Cognitive Impairment or Early Stages of Dementia and Their Caregivers: Cross-Sectional Study. J Med Internet Res. 2020 Jun 1;22(6):e17253. doi: 10.2196/17253. PMID 32442136
- [Derived] Anderberg P, Barnestein-Fonseca P, Guzman-Parra J, Garolera M, Quintana M, Mayoral-Cleries F, Lemmens E, Sanmartin Berglund J. The Effects of the Digital Platform Support Monitoring and Reminder Technology for Mild Dementia (SMART4MD) for People With Mild Cognitive Impairment and Their Informal Carers: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2019 Jun 21;8(6):e13711. doi: 10.2196/13711. PMID 31228177